CLINICAL TRIAL: NCT03512184
Title: The YMCA's Diabetes Prevention Program (YMCA's DPP) for the Treatment of Nonalcoholic Fatty Liver Disease
Brief Title: YMCA Diabetes Prevention Program for the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: YMCA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1709018542
Record Dates: First submitted 2018-02-06; First posted 2018-04-30 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Weight Loss; NAFLD; Liver Diseases
MeSH Terms: conditions — Weight Loss; Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YMCA Class (Other): This Arm's objective is to determine the effect of the YMCA's Diabetes Prevention Program on NAFLD as determined by comparison of liver enzymes pre- and post- program.
  Interventions: Behavioral: YMCA class

INTERVENTIONS:
Behavioral: YMCA class — The Gastroenterologists of Weill Cornell Medical College that are associated with this trial want to implement the YMCA's DPP in the NAFLD population as a structured lifestyle modification/educational intervention. The hypothesis is that the NAFLD patients who complete the YMCA's DPP will also have weight loss and improvement in hepatic steatosis. Importantly, positive results in this New York City-based pilot study would provide a strong rationale for determining whether such a program could be useful to treat NAFLD at established YMCA DPP sites across the country.

SUMMARY:
This study is for men and women have been diagnosed with non-alcoholic fatty liver disease (NAFLD) and will consequently participate in the YMCA's Diabetes Prevention Program.

DETAILED DESCRIPTION:
This study is for men and women who participate in the YMCA's Diabetes Prevention Program (YMCA's DPP) and have been diagnosed with non-alcoholic fatty liver disease (NAFLD). There will be no administration of study drug. The purpose of this study is to see if participation in the YMCA's DPP will result in weight loss and improvement in the liver in patients with fatty liver disease.

Eligible participants will visit Weill Cornell Medical College's Gastroenterology and Hepatology clinic to review their medical history, physical examination, complete a survey, and conduct imaging tests (FibroScan, ultrasound, DEXA scan) for their baseline visit. Blood will be collected as part of standard practice. An additional blood sample will be collected for storage. Subjects will complete 9 out of 16 weekly sessions. The YMCA's program will be conducted at Weill Cornell Medical College Gastroenterology and Hepatology Division.

Participants will be in the YMCA program for about 1 year and an additional 1 year in the long-term follow-up for data collection.

Participants will be compensated for their time.

Key eligibility criteria:

1. Men and women over 18 years of age.
2. Diagnosed with Non-alcoholic Fatty liver disease.
3. Detailed eligibility reviewed when contacting the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Must provide signed written informed consent and agree to comply with the study protocol
3. BMI >25 kg/m²
4. Hepatic steatosis by imaging or histology
5. Baseline Fibroscan CAP score > 238 dB/m
6. ALT >19IU/mL in females, ALT >30IU/mL in males

Exclusion Criteria:

1. Unclear etiology of liver disease
2. Competing etiologies for hepatic steatosis
3. Co-existing causes of chronic liver disease according to standard diagnostic testing including, but not restricted to:

   * Positive hepatitis B surface antigen
   * Positive hepatitis C virus RNA
   * Suspicion of drug-induced liver disease
   * Alcoholic liver disease
   * Autoimmune hepatitis
   * Wilson's disease
   * Hemochromatosis
   * Primary biliary cholangitis or primary sclerosing cholangitis
4. Known or suspected hepatocellular carcinoma
5. Current or recent history (<5 years) of significant alcohol consumption. For men, significant consumption is defined as >30g of alcohol per day. For women, it is defined as >20g of alcohol per day.
6. Compensated and decompensated cirrhosis (clinical and/or histologic evidence of cirrhosis). NASH patients with fibrosis stage = 4 according to the NASH CRN fibrosis staging system are excluded.
7. Pregnant females
8. Mental instability or incompetence, such that the validity of the informed consent or ability to be compliant with the study is uncertain
9. Inability to perform Fibroscan and/or invalid study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Effect of the YMCA's Diabetes Prevention Program on NAFLD | 104 weeks from the start of the study
  Determine the effect of the YMCA's Diabetes Prevention Program on NAFLD as determined by comparison of liver enzymes pre- and post- program - we'll look at the changes of ALT levels to determine the aforementioned. We will perform these diagnostic tests in order to determine the effectiveness of the 16 weeks of sessions.
Determine if Liver Fat via Fibroscan Controlled Attentuation Pattern score has decreased as a result of YMCA program | 104 weeks from the start of the study
  Evaluate the amount of liver fat as determined by Fibroscan Controlled Attenuation Pattern (CAP) score in patients with NAFLD pre- and post- participation in the diabetes prevention program with the YMCA. The CAP range should be 100-400, without any sub-scales reported. Lower values in the range represent less 'fat', making it a better score.

SECONDARY OUTCOMES:
Measuring the effectiveness of the YMCA Program, as per SF-36 patient-reported questionnaires | 104 weeks from the start of the study
  Determine the effect of YMCA's DPP on quality of life in patients with NAFLD as per SF-36 questionnaire.
Measuring the effectiveness of the YMCA Program, as per each patient's BMI | 104 weeks from the start of the study
  Determine the effect of YMCA's DPP on BMI in patients with NAFLD. We are reporting this as an aggregate of Body Mass Index.
Measuring the effectiveness of the YMCA Program, as per the DEXA scan | 104 weeks from the start of the study
  Determine the effect of YMCA's DPP on body composition (aggregated via body fat percentage and lean and fat body mass) using dual-energy X-ray absorptiometry (DEXA).
Measuring the effectiveness of the YMCA Program, as per metabolic blood work that's analyzed | 104 weeks from the start of the study
  Determine the effect of YMCA's DPP on levels of systemic factors linked to the metabolic syndrome. The metabolites that will be studied are all research-related blood work.

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Kumar, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided